CLINICAL TRIAL: NCT03646305
Title: Singing Your Negative Body-Related Thoughts: A Randomized Controlled Trial of a New Cognitive Defusion Strategy
Brief Title: Singing Your Negative Body-Related Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Mills, Professor, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-111
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Body Dissatisfaction

STUDY DESIGN:
Intervention Model Description: This was a single-center, parallel-group study with balanced randomization of participants into four conditions; two experimental and two control [1:1:1:1]. This is a non-inferiority study to examine whether singing is as effective as verbal repetition as a cognitive defusion strategy for body image distress.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Verbally repeat body-related thoughts (Experimental): A cognitive defusion strategy in which participants repeat a target unwanted thought out loud and as quickly as possible for 60 seconds.
  Interventions: Behavioral: Cognitive Defusion
- Sing negative body-related thoughts (Experimental): A cognitive defusion strategy in which participants sing a target unwanted thought to the tune of 'twinkle, twinkle' for 60 seconds
  Interventions: Behavioral: Cognitive Defusion
- Verbally repeat body-unrelated thoughts (No Intervention): A control condition in which participants repeat the phrase "I am talking" out loud and as quickly as possible for 60 seconds.
- Sing body-unrelated thoughts (No Intervention): A control condition in which participants sing the phrase "I am singing" to the tune of 'twinkle, twinkle' for 60 seconds

INTERVENTIONS:
Behavioral: Cognitive Defusion — Cognitive defusion aims to change one's relationship to their thoughts - as opposed to changing the content, form, or frequency - by reframing internal experiences as less threatening (Hayes, Luoma, Bond, Masuda, & Lillis, 2006). It is the process of detaching the link between one's thoughts and perceptions of reality and acknowledging the role one's thoughts play in their internal events. A number of techniques have been developed to remove the literal quality of such thoughts, including repeating the thought, and, more recently, singing the thought.
  Arms: Sing negative body-related thoughts; Verbally repeat body-related thoughts

SUMMARY:
Study Objectives:

1. Examine whether singing can be used as a cognitive defusion strategy to change one's appraisals of body-related thoughts so they are less threatening to the individual.
2. Explore whether this technique can change the appraisals of one's body (i.e. increasing body satisfaction, increasing body esteem, decreasing the drive towards thinness), as well as increase mood and self-esteem.
3. Compare singing to the defusion strategy of verbal repetition, as well as control conditions, to determine the effectiveness of these techniques.
4. Examine whether defusion techniques would be particularly beneficial for individuals with high thought-shape fusion

Study Hypotheses:

The primary hypothesis was that the cognitive defusion conditions, namely verbal repetition and singing, would foster greater detachment (i.e. defusion) from negative body-related thoughts and change thought appraisals such that these thoughts were less believable and less negative, and the individual was more willing, less likely to avoid, and less uncomfortable when engaging with these thoughts than the control conditions.

Secondary hypotheses propose that these defusion techniques will reduce negative body-related cognitions such as body image distress, drive for thinness, and body dissatisfaction to a greater extent than the control conditions. Moreover, compared to the control condition, these techniques are expected to be superior in reducing negative mood and improving self-esteem. Finally, better outcomes are expected from those in the defusion conditions who practice the technique as instructed (i.e. better homework adherence). Due to the novelty of this intervention, no specific hypotheses have been made regarding whether singing will equal or differ from verbal repetition on the aforementioned outcome measures. Moreover, due to the exploratory nature of applying defusion techniques with individuals with thought-shape fusion, no specific hypotheses have been made around anticipated changes in the perception of the thought, body image satisfaction, mood, self-esteem, and cognitive defusion within this population.

DETAILED DESCRIPTION:
Eating disorders are characterized by intense mental preoccupation with body shape and weight. Even in the absence of disordered eating, high levels of body dissatisfaction prospectively predict depression and low self-esteem in young women. Common intervention strategies, such as challenging the validity of negative body-related thoughts, often have limited success. Recent research suggests that accepting, rather than challenging, negative body-related thoughts may reduce body image distress by changing the relationship with those thoughts. For example, continually repeating or even singing an unwanted thought has been shown to reduce the believability and discomfort associated with that thought, through a technique known as cognitive defusion. The current study aims to extend the literature on cognitive defusion and test its effectiveness in the treatment of body dissatisfaction. In a randomized controlled trial design, 122 female restrained eaters were randomly assigned to practice either 1) verbally repeating negative body-related thoughts, 2) singing negative body-related thoughts, 3) verbally repeating body-unrelated thoughts (control), or 4) singing body-unrelated thoughts (control). The goal of this study was to determine whether singing one's negative body-related thoughts could lead to greater changes in perception of the thought, body image satisfaction, mood, and self-esteem relative to a control condition when practiced twice daily for one week.

ELIGIBILITY:
Inclusion Criteria:

* Restrained eaters, as indicated by a score of 15 or greater on the Revised Restraint Scale (Polivy, Herman, & Howard, 1988)
* Identify as female
* Age 17 and older

Exclusion Criteria:

* Under age 17
* Do not identify as female
* Scores below 15 on the Revised Restraint Scale (Polivy, Herman, & Howard, 1988).

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keisha C Gobin, BA, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Polivy, J., Herman, P. H., & Howard, K. I. (1988). Restraint scale: Assessment of dieting. In M. Hersen & A. S. Bel lack (Eds.), Dictionary of behavioral assessment techniques (pp. 377- 380). Elmsford, NY: Pergamon Press.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Undergraduate Research Participant Pool of students enrolled in Introduction to Psychology at York University. Participants were individuals who reported restrained eating behaviours and attitudes as determined by an eligibility screener conducted online at the start of the academic year (September 2018).
Pre-assignment Details: All participants who were enrolled in this study were assigned to a condition.
Period: Overall Study
Arm/Group | Verbally Repeat Body-related Thoughts | Sing Negative Body-related Thoughts | Verbally Repeat Body-unrelated Thoughts | Sing Body-unrelated Thoughts
Started | 32 | 35 | 33 | 33
Received Treatment | 31 | 35 | 32 | 32
No Treatment Recieved | 1 | 0 | 1 | 1
Completed | 27 | 33 | 31 | 31
Not Completed | 5 | 2 | 2 | 2
Not completed — Lost to Follow-up | 4 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verbally Repeat Body-related Thoughts | Sing Negative Body-related Thoughts | Verbally Repeat Body-unrelated Thoughts | Sing Body-unrelated Thoughts | Total
Number analyzed (Participants) | 32 | 35 | 33 | 33 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.70 (6.10) | 20.49 (3.42) | 19.66 (1.75) | 22.66 (7.22) | 20.87 (5.11)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Only females were recruited for this study
  Participants
    Female | 32 | 35 | 33 | 33 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Arab/West Asian | 7 | 13 | 5 | 5 | 30
  Race/Ethnicity: Black | 2 | 2 | 2 | 0 | 6
  Race/Ethnicity: East Asian | 2 | 4 | 2 | 2 | 10
  Race/Ethnicity: Latin American | 2 | 0 | 1 | 1 | 4
  Race/Ethnicity: South Asian | 5 | 3 | 3 | 6 | 17
  Race/Ethnicity: South East Asian | 2 | 0 | 2 | 2 | 6
  Race/Ethnicity: White | 9 | 11 | 10 | 12 | 42
  Race/Ethnicity: Mixed | 2 | 1 | 4 | 1 | 8
  Race/Ethnicity: Other | 0 | 1 | 3 | 2 | 6
  Race/Ethnicity: Declined to response | 1 | 0 | 1 | 2 | 4
Restrained Eating [Mean (Standard Deviation); unit: units on a scale] — The Revised Restraint Scale is a 10-item measure of restrained eating behaviours and attitudes. Participants rate statements about themselves on a Likert scale ranging from 0 to 3 or 0 to 4. A score of 15 or higher is indicative of restrained eating. Total score can range from 0 to 35.
  units on a scale | 21.65 (4.27) | 19.55 (4.15) | 23.27 (4.06) | 20.68 (3.20) | 21.23 (4.12)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was collected at the end of visit two but is included as a baseline measure. BMI was not collected at the start because many subjects ask to know their weight, which can influence their behaviours/self-reports. Data from participants who dropped out is not included. Population: BMI was not collected from participants who dropped out.
  kg/m^2
    number analyzed (Participants) | 27 | 33 | 31 | 31 | 122
    (all) | 26.17 (6.41) | 24.79 (6.20) | 26.89 (5.63) | 24.59 (4.27) | 25.59 (5.69)

OUTCOME MEASURES:

1. Primary Outcome: Self-Ratings of Thought Appraisals (Believability)
Description: Participants rated the believability of their body-related thought on a visual analogue scale that ranges from 0-100. Higher scores means greater believability of this negative thought.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Verbally Repeat Body-related Thoughts | Sing Negative Body-related Thoughts | Verbally Repeat Body-unrelated Thoughts | Sing Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 78.33 (24.01) | 77.97 (25.47) | 83.23 (19.97) | 74.74 (22.42)
  Post-intervention | 61.56 (29.93) | 62.09 (27.80) | 65.90 (25.01) | 55.23 (31.88)
  Follow-up | 53.11 (33.44) | 46.94 (28.15) | 53.68 (27.02) | 45.52 (26.30)
Statistical Analysis 1: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental,control) × 2(Activity: singing,verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, believability of thought were equivalent across time; Test type: Non-Inferiority — This was a single-center, parallel-group study with balanced randomization of participants into one of four conditions. Condition (experimental: body-related thoughts vs control: neutral thoughts) was fully crossed with technique (singing vs verbal repetition) . This was a non-inferiority study to primarily examine whether singing is as effective as verbal repetition as a cognitive defusion strategy for body image distress; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; A paired sample t-test was conducted to measure differences in believability of thought from baseline to post-intervention. Null hypothesis: there would be no significant difference in believability of thought from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; A paired sample t-test was conducted to measure differences from post-intervention to follow-up. Null hypothesis: there would be no significant differences in believability of thought from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal believability scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal believability scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in believability scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions have equivalent believability scores across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on believability scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no significant difference between 4 conditions on believability; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

2. Primary Outcome: Self-Ratings of Thought Appraisals (Negativity)
Description: Participants rated the negativity of their body-related thought on a visual analogue scale that ranges from 0-100. Higher scores means that the negative thought is perceived to be more negative.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-Up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Verbally Repeat Body-related Thoughts | Sing Negative Body-related Thoughts | Verbally Repeat Body-unrelated Thoughts | Sing Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 68.96 (29.04) | 75.39 (28.22) | 71.61 (28.07) | 71.90 (27.67)
  Post-intervention | 70.93 (28.22) | 68.64 (32.30) | 66.06 (31.26) | 59.90 (33.99)
  Follow-up | 66.78 (30.52) | 65.88 (32.21) | 48.58 (34.00) | 47.74 (33.38)
Statistical Analysis 1: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, appraisal of target thought were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.005, ANOVA
Statistical Analysis 3: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in negativity from baseline to post-intervention. Null hypothesis: the control conditions would have no significant difference in negativity from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.002, t-test, 2 sided
Statistical Analysis 4: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in negativity from post-intervention to follow-up. Null hypothesis: the control conditions would have no significant difference in negativity from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; A paired sample t-test was conducted to measure differences in negativity from baseline to post-intervention. Null hypothesis: there would be no significant difference in negativity scores from baseline to post-intervention in the experimental conditions; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.025, t-test, 2 sided
Statistical Analysis 6: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in negativity from post-intervention to follow-up. Null hypothesis: the experimental conditions would have no significant difference in negativity scores from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.025, t-test, 2 sided
Statistical Analysis 7: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal negativity scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal negativity scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in negativity scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 10: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on negativity scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 11: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between four conditions on negativity scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

3. Primary Outcome: Self-Ratings of Thought Appraisals (Discomfort)
Description: Participants rated the discomfort of their body-related thought on a visual analogue scale that ranges from 0-100. Higher scores means that the thought is perceived to be more uncomfortable.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 33 | 27 | 31 | 31
score on a scale
  Baseline | 79.97 (20.73) | 63.48 (33.62) | 74.06 (28.61) | 69.90 (31.77)
  Post-intervention | 59.48 (28.55) | 54.93 (37.19) | 53.42 (33.49) | 54.42 (31.75)
  Follow-up | 51.45 (29.84) | 46.85 (35.20) | 42.74 (34.06) | 41.61 (29.96)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at p< .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, levels of discomfort were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in levels of discomfort from baseline to post-intervention. Null hypothesis: there would have no significant differences in discomfort levels from baseline to post-intervention across samples; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in levels of discomfort from post-intervention to follow-up. Null hypothesis: there would be no significant differences in discomfort levels from post-intervention to follow-up across samples; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of discomfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal levels of discomfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in levels of discomfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in levels of discomfort across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on levels of discomfort; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no significant difference between 4 conditions on discomfort levels; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

4. Primary Outcome: Self-Ratings of Thought Appraisals (Willingness)
Description: Participants rated their willingness to have their body-related thought on a visual analogue scale that ranges from 0-100. Higher scores means that they are more willing to have the thought.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 61.03 (28.05) | 62.41 (30.87) | 65.74 (29.83) | 60.90 (23.29)
  Post-intervention | 52.58 (31.49) | 55.15 (31.04) | 53.55 (33.72) | 58.42 (24.10)
  Follow-up | 55.15 (30.54) | 50.22 (30.92) | 45.10 (29.24) | 48.39 (30.94)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, willingness to engage with target thought were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in willingness to engage with target thought from baseline to post-intervention. Null hypothesis: there would be no difference in willingness scores from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in willingness to engage with target thought from post-intervention to follow-up. Null hypothesis: there would be no significant difference in willingness scores from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.053, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal willingness scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal willingness to engage with the target thought; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all 4 conditions were equivalent in willingness to engage; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in willingness to engage with the target thought across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on willingness to engage; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between 4 conditions on willingness to engage; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

5. Primary Outcome: Self-Ratings of Thought Appraisals (Avoidance)
Description: Participants rated their avoidance of their body-related thought on a visual analogue scale that ranges from 0-100. Higher scores means greater avoidance of the thought.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 59.39 (35.30) | 50.63 (34.73) | 44.52 (32.93) | 51.81 (32.95)
  Post-intervention | 53.42 (34.13) | 52.11 (36.92) | 46.45 (33.41) | 45.52 (32.50)
  Follow-up | 56.45 (32.38) | 39.07 (32.97) | 36.87 (32.38) | 36.48 (32.14)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, avoidance of target thought were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in avoidance of target thought from baseline to post-intervention. Null hypothesis: there would be no significant differences in avoidance from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in avoidance of target thought from post-intervention to follow-up. Null hypothesis: there would be no significant differences in avoidance from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would show equal avoidance of target thought; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal avoidance of target thought; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all 4 conditions were equivalent in avoidance of target thought; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in avoidance of target thought across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on avoidance of target thought; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between 4 conditions on avoidance of target thought; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

6. Primary Outcome: Self-Ratings of Cognitive Fusion (Cognitive Fusion Questionnaire)
Description: The Cognitive Fusion Questionnaire includes 7 items measured on a 7 item Likert scale and will be used to measure changes in cognitive fusion. Higher scores indicate higher degree of cognitive fusion. Total scores can range from 7 to 49.
Time Frame: Baseline and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Verbally Repeat Body-related Thoughts | Sing Negative Body-related Thoughts | Verbally Repeat Body-unrelated Thoughts | Sing Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 36.56 (9.55) | 32.52 (10.59) | 33.65 (9.03) | 31.52 (11.17)
  Follow-Up | 33.30 (10.84) | 32.91 (10.19) | 32.65 (10.85) | 29.97 (9.94)
Statistical Analysis 1: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, cognitive delusion were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of cognitive defusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal levels of cognitive defusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in levels of cognitive defusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in levels of cognitive defusion across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance alpha level .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on levels of cognitive defusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Verbally Repeat Body-related Thoughts vs Sing Negative Body-related Thoughts vs Verbally Repeat Body-unrelated Thoughts vs Sing Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance alpha level .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between four conditions on levels of cognitive defusion; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

7. Secondary Outcome: Self-Ratings of Body Image Cognitions (Weight Dissatisfaction)
Description: Participants rated their weight dissatisfaction on a visual analogue scale that ranges from 0-100. Higher scores means greater weight dissatisfaction.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 33 | 27 | 31 | 31
score on a scale
  Baseline | 59.15 (31.28) | 71.22 (29.22) | 66.10 (33.09) | 68.68 (29.11)
  Post-intervention | 51.70 (28.13) | 62.33 (30.05) | 50.81 (33.03) | 58.81 (32.07)
  Follow-Up | 49.64 (27.52) | 52.85 (32.04) | 45.39 (30.52) | 50.45 (26.84)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, weight dissatisfaction were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in weight dissatisfaction from baseline to post-intervention. Null hypothesis: there would be no significant differences in weight dissatisfaction from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; A paired sample t-test was conducted to measure differences in weight dissatisfaction from post-intervention to follow-up. Null: there would be no differences in weight dissatisfaction from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal weight dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal weight dissatisfaction scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA used to analyze Intervention x Activity interaction. Null: On average, all 4 conditions were equivalent in weight dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in weight dissatisfaction across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on weight dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between four conditions on weight dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

8. Secondary Outcome: Self-Ratings of Body Image Cognitions (Appearance Dissatisfaction)
Description: Participants rated their appearance dissatisfaction on a visual analogue scale that ranges from 0-100. Higher scores means greater appearance dissatisfaction.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 55.18 (31.77) | 58.67 (33.63) | 47.55 (31.88) | 50.90 (32.90)
  Post-intervention | 51.24 (28.79) | 57.67 (31.12) | 50.26 (29.00) | 50.87 (33.27)
  Follow-up | 51.03 (27.01) | 46.41 (30.78) | 35.26 (28.47) | 44.81 (24.46)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, appearance dissatisfaction were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in appearance dissatisfaction from baseline to post-intervention. Null hypothesis: the control conditions would have no significant difference in appearance dissatisfaction from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in appearance dissatisfaction from post-intervention to follow-up. Null hypothesis: the control conditions would have no significant difference in appearance dissatisfaction from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal appearance dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal appearance dissatisfaction scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in appearance dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in appearance dissatisfaction across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on appearance dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between four conditions on appearance dissatisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

9. Secondary Outcome: Self-ratings of Body Image Distress (Body Image State Scale)
Description: The Body Image State Scale was used as part of a standard questionnaire package to measure changes in body image cognitions. Participants rated 6 items on a 9-point Likert scale ranging from 1 to 9, for a possible total score of 6 to 54, with higher scores indicating greater body image satisfaction (i.e. positive body image).
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 33 | 27 | 31 | 31
score on a scale
  Baseline | 26.64 (8.38) | 25.44 (9.12) | 25.71 (8.25) | 24.74 (8.75)
  Post-intervention | 27.82 (9.35) | 26.41 (9.60) | 27.81 (8.96) | 26.32 (7.56)
  Follow-up | 29.12 (10.28) | 28.19 (10.96) | 30.61 (8.75) | 30.48 (9.38)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, body state image satisfaction were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; A paired sample t-test was conducted to measure the difference in state body image satisfaction from baseline to post intervention. Null hypothesis: there would be no significant differences in state body image satisfaction from baseline to post intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; A paired sample t-test was conducted to measure the difference in state body image satisfaction from post intervention to follow-up. Null hypothesis: there would be no significant differences in state body image satisfaction from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal body state image satisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal state body satisfaction scores; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in state body image satisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in state body image satisfaction across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance alpha level .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on state body image satisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance alpha level.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between four conditions on state body image satisfaction; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

10. Secondary Outcome: Self-Ratings of Mood (Anxiety)
Description: Participants rated their anxiety on a visual analogue scale that ranges from 0-100. Higher scores means greater anxiety.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 33 | 27 | 31 | 31
score on a scale
  Baseline | 51.45 (31.39) | 49.15 (30.14) | 37.94 (28.87) | 52.68 (24.44)
  Post-intervention | 43.55 (30.08) | 32.67 (28.25) | 27.68 (27.83) | 39.65 (27.81)
  Follow-up | 41.48 (29.81) | 35.33 (26.28) | 26.74 (26.78) | 37.61 (26.47)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, state body image satisfaction were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; A paired sample t-test was conducted to measure differences in anxious mood from baseline to post-intervention. Null hypothesis: there would be no significant difference in anxious mood from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in anxious mood from post-intervention to follow-up. Null hypothesis: there would be no significant difference in anxious mood from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of anxiety; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal levels of anxiety; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in levels of anxiety; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in levels of anxiety across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on levels of anxiety; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between the four conditions on levels of anxiety; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

11. Secondary Outcome: Self-Ratings of Mood (Depression)
Description: Participants rated their depressive mood on a visual analogue scale that ranges from 0-100. Higher scores means greater depressive mood.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 30.76 (30.93) | 27.85 (28.52) | 25.52 (25.88) | 36.94 (29.77)
  Post-intervention | 27.12 (30.57) | 21.67 (25.26) | 19.55 (25.18) | 23.84 (25.07)
  Follow-up | 26.82 (29.00) | 25.96 (28.61) | 19.74 (24.46) | 27.65 (22.76)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, levels of depressive mood were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in depressive mood from depressive mood from baseline to post-intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in depressive mood from post-intervention to follow-up. Null hypothesis: there would be no significant differences in depressive mood from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of depressive mood; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal levels of depressive mood; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in levels of depressive mood; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in levels of depressive mood across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on levels of depressive mood; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 9: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no difference between 4 conditions on levels of depressive mood; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

12. Secondary Outcome: Self-Ratings of Mood (Happiness)
Description: Participants rated their happiness on a visual analogue scale that ranges from 0-100. Higher scores means greater happy mood.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 57.85 (24.68) | 54.59 (24.10) | 52.00 (25.15) | 51.45 (21.81)
  Post-intervention | 50.15 (30.82) | 53.63 (26.47) | 57.58 (29.56) | 55.84 (25.64)
  Follow-up | 50.03 (26.98) | 49.78 (29.54) | 55.35 (22.72) | 49.06 (25.36)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, levels of happiness were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of happiness; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would have equal levels of happiness; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in levels of happiness; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in levels of happiness across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on levels of happiness; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no differences between four conditions on levels of happiness; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

13. Secondary Outcome: Self-Ratings of Mood (Confidence)
Description: Participants rated their confidence on a visual analogue scale that ranges from 0-100. Higher scores means greater confidence.
Time Frame: Baseline, Post-Intervention (Day 1), and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 27 | 33 | 31 | 31
score on a scale
  Baseline | 48.91 (26.37) | 40.52 (25.38) | 47.77 (29.97) | 42.03 (22.61)
  Post-intervention | 42.12 (31.34) | 37.30 (25.72) | 52.39 (32.67) | 45.26 (25.95)
  Follow-up | 46.88 (26.14) | 43.81 (25.87) | 50.26 (28.09) | 47.39 (27.09)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, levels of confidence were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of confidence; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal levels of confidence; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA was used to analyze Intervention x Activity interaction. Null: On average, all four conditions were equivalent in levels of confidence; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions are equivalent in levels of confidence across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; [analysis description as in outcome 12, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; [analysis description as in outcome 12, analysis 7]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

14. Secondary Outcome: Self-Ratings of Self-Esteem (State Self Esteem Scale)
Description: The State Self Esteem Scale is a 20-item measure used to assess changes in state self esteem, rated on a 5-point Likert scale. Total scores can range from 5 to 100. Higher scores indicate higher self-esteem.
Time Frame: Baseline and Follow-up (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 33 | 27 | 31 | 31
score on a scale
  Baseline | 62.36 (15.60) | 58.26 (15.73) | 59.65 (17.15) | 58.58 (13.90)
  Follow-up | 64.52 (16.30) | 61.96 (14.13) | 65.58 (16.24) | 62.97 (15.48)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to measure main effect of time. Null: Across the sample, level of self-esteem were equivalent across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Paired sample t-tests was conducted to measure differences in self-esteem from post-intervention to follow-up. Null hypothesis: there would be no significant differences in self-esteem from post-intervention to follow-up; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Intervention. Null: On average, the experimental conditions and control conditions would have equal levels of self-esteem; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze main effect of Activity. Null: On average, singing and verbal repetition would result in equal levels of self-esteem; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; Twenty-eight participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post-intervention, follow-up) mixed ANOVA used to analyze Intervention x Activity interaction. Null: On average, all four conditions have equivalent levels of self-esteem; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect a moderate effect size (.25) at a significance level of alpha .05 in a mixed ANOVA according to a power analysis using GPower 3.1. A 2 (Intervention: experimental, control) × 3 (Time: baseline, post-intervention, follow-up) mixed ANOVA was used to measure Time x Intervention interactions. Null: experimental and control conditions have equivalent levels of self-esteem across time; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Activity interaction. Null: Across time, there would be no difference between singing and verbal repetition on levels of self-esteem; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; 28 participants per condition (N=112) would provide sufficient power (0.8) to detect moderate effect size (.25) at significance level of alpha.05 in mixed ANOVA according to power analysis using GPower 3.1. A 2(Intervention: experimental, control) × 2(Activity: singing, verbal repetition) × 3(Time: baseline, post, follow-up) mixed ANOVA was used to analyze Time x Intervention x Activity interaction. Null: Across time, there would be no differences between four conditions on levels of self-esteem; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

15. Secondary Outcome: Self-Rating of Homework Adherence (Homework Adherence Questionnaire)
Description: Homework adherence was determined by the total number of seconds spent practicing the defusion technique over the course of the week. There is no total scale range available for this measure.
Time Frame: Homework completion across seven days (14 time points)
Population: Many homework log entries were missing due to failure to return the forms, forgetting to fill out the form, or not practicing. As such, 61 of 122 participants provided enough data to be included in this homework compliance analysis.
Measure: Mean (Standard Deviation); unit: seconds per week
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 12 | 13 | 16 | 20
seconds per week | 32.64 (8.25) | 29.79 (1.07) | 29.81 (1.43) | 32.24 (6.10)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; All mediation analyses were conducted using the PROCESS SPSS macro version 3.2 (Hayes, 2018). We tested model 4, which includes one outcome variable, one predictor, one mediator, and room for covariates. We examined the meditational effect of homework adherence on the relationship between intervention and each outcome measure. Null: homework adherence does not mediate any relationships between intervention condition and outcome measures; Test type: Other — Mediation Analysis that examined whether greater homework adherence strengthened the relationship between condition and outcome; p > 0.05, Mediation Analyses
Statistical Analysis 2: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; All mediation analyses were conducted using the PROCESS SPSS macro version 3.2 (Hayes, 2018). We tested model 4, which includes one outcome variable, one predictor, one mediator, and room for covariates. We examined the meditational effect of homework adherence on the relationship between activity and each outcome measure. Null: homework adherence does not mediate any relationships between activity condition and outcome measures; Test type: Other — [test comment as in outcome 15, analysis 1]; p > 0.05, Mediation Analyses

16. Secondary Outcome: Self-Rating of Thought-Shape Fusion (Thought-Shape Fusion Questionnaire)
Description: The Thought-Shape Fusion Questionnaire was used to assess the extent to which thinking about a forbidden food or behaviour produces a change in one's perception of their body shape and weight. It is a 34-item measure that asks participants to rate how well an item describes them on a 5 point Likert scale from 0 to 4. Total scores can range from 0 to 136, with higher scores indicating greater fusion to body- or food-related thoughts.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sing Negative Body-related Thoughts | Verbally Repeat Body-related Thoughts | Sing Body-unrelated Thoughts | Verbally Repeat Body-unrelated Thoughts
Number analyzed (Participants) | 33 | 27 | 31 | 31
score on a scale | 43.67 (37.70) | 45.56 (39.79) | 32.77 (29.94) | 35.65 (26.18)
Statistical Analysis 1: Comparison: Sing Negative Body-related Thoughts vs Verbally Repeat Body-related Thoughts vs Sing Body-unrelated Thoughts vs Verbally Repeat Body-unrelated Thoughts; All moderation analyses were conducted using the PROCESS SPSS macro version 3.2 (Hayes, 2018). We tested model 1, which includes one outcome variable, one predictor, and one moderator. Thought-shape fusion was examined as a potential moderator of the relationship between intervention condition and outcome measures. Null: thought-shape fusion does not significantly moderate the relationship between intervention condition and state self-esteem; Test type: Other — Thought-shape fusion was examined as a potential moderator of the relationship between intervention condition and outcome measures; p < 0.001, Moderation Analyses — No other outcome measure was moderated by thought-shape fusion scores

ADVERSE EVENTS:
Time Frame: Participants were given the opportunity to withdraw at any point during the study and were monitored for adverse events throughout the completion of the study (ie. day 1 to day 7).
Arm/Group | Verbally Repeat Body-related Thoughts | Sing Negative Body-related Thoughts | Verbally Repeat Body-unrelated Thoughts | Sing Body-unrelated Thoughts
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/33 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/33 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/27 | 0/33 | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
No limitations or caveats to declare

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03646305/Prot_SAP_000.pdf